CLINICAL TRIAL: NCT03239262
Title: Assessment of the Effect of Left Atrial Cryoablation Enhanced by Ganglionated Plexi Ablation in the Treatment of Atrial Fibrillation in Patients Undergoing Open Heart Surgery
Brief Title: Left Atrial Cryoablation Enhanced by Ganglionated Plexi Ablation in the Treatment of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-Cardiosurgery-1
Record Dates: First submitted 2017-07-26; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Mitral Valve Disease; Coronary Artery Disease; Tricuspid Valve Disease; Aortic Valve Disease; Atrial Fibrillation
Keywords: Atrial Fibrillation; Left Atrial Cryoablation; Ganglionated Plexi; Open-Heart Surgery
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease; Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Two groups of patients undergoing standard treatment have been compared retrospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group GP (Experimental): Thirty-five patients (35%) from our population underwent concomitant mapping and radiofrequency ablation of ganglionated plexi (Group GP).
  Interventions: Procedure: Concomitant Mapping and Radiofrequency Ablation
- Group LA (Experimental): Sixty five patients (65%) in whom no intervention related to ganglionated plexi was performed (Group LA).
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: Concomitant Mapping and Radiofrequency Ablation — Mapping of GP around the orifice of pulmonary veins was performed, together with their radiofrequency ablation. In the area of right-side pulmonary veins, the procedure was performed prior to initiation of extracorporeal circulation. In case of the left-side PVs; the procedure was performed after initiation of extracorporeal circulation. Part of this procedure was also a decision and ablation of the ligament of Marshall.
  GP mapping was performed using high-frequency stimulation (1000 beats min-¹, potential 18V, pulse width 1.5ms). The indication for GP ablation was a doubling in the R-R interval in the sinus rhythm, or ventricular rate slowing of more that 50% associated with a decrease of blood pressure>20mmHg in patients with AF. In case of a positive response, radiofrequency ablation of the ganglia was performed following switching of the pen at the console. This procedure was repeated until the activity of the ganglia has disappeared.
  Arms: Group GP
Procedure: No intervention — No intervention was performed in patients without ganglionated plexi.
  Arms: Group LA

SUMMARY:
The aim of our study was to investigate, whether enhancement of left atrial cryoablation by ablation of the autonomic nervous system of left atrium leads to influencing the outcomes of surgical treatment of atrial fibrillation in patients with structural heart disease undergoing open-heart surgery.

DETAILED DESCRIPTION:
The observed patient file consisted of 100 patients, who have undergone a combined open-heart surgery at our department between July 2012 and December 2014. The patients were indicated for the surgical procedure due to structural heart disease, and suffered from paroxysmal, persistent, or long-standing persistent atrial fibrillation. In all cases, left atrial cryoablation was performed in the extent of isolation of pulmonary veins, box lesion, connecting lesion with mitral annulus, amputation of the left atrial appendage and connecting lesion of the appendage base with left pulmonary veins. Furthermore, thirty-five of the patients underwent mapping and radiofrequency ablation of ganglionated plexi, together with decision and ablation of the ligament of Marshall.

ELIGIBILITY:
Inclusion Criteria:

* Indication for open-heart surgery (mitral valve disease and/or tricuspidal valve disease and/or aortic valve disease and/or coronary artery disease and/or other)
* Concomitant paroxysmal, persistent, long standing persistent atrial fibrillation
* Signing of the informed consent

Exclusion Criteria:

* Age below 40 and over 80 years of age
* Left ventricular ejection fraction below 25%
* Left atrium diameter over 60mm
* Permanent atrial fibrillation
* Polymorbidity (Euroscore II over 10)
* Emergency surgery
* Renal insufficiency (creatinine over 200 umol/l)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Sinus Rhythm | 30 months
  The primary outcome was establishment and duration of sinus rhythm in the course of one-year follow-up.

SECONDARY OUTCOMES:
Recurrence of Atrial Fibrillation and the Presence of a Mitral Valve Surgery | 30 months
  The secondary outcome was the detection of relationship between the recurrence of atrial fibrillation and the presence of a mitral valve surgery, the presence of a mitral and tricuspid valves surgery and the left atrium diameter >50 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Barta, MD, Principal Investigator — University Hospital Ostrava; Radim Brat, MD,PhD,MBA, Study Chair — University Hospital Ostrava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hou Y, Scherlag BJ, Lin J, Zhang Y, Lu Z, Truong K, Patterson E, Lazzara R, Jackman WM, Po SS. Ganglionated plexi modulate extrinsic cardiac autonomic nerve input: effects on sinus rate, atrioventricular conduction, refractoriness, and inducibility of atrial fibrillation. J Am Coll Cardiol. 2007 Jul 3;50(1):61-8. doi: 10.1016/j.jacc.2007.02.066. Epub 2007 Jun 18. PMID 17601547
- [Background] Katritsis DG, Giazitzoglou E, Zografos T, Pokushalov E, Po SS, Camm AJ. Rapid pulmonary vein isolation combined with autonomic ganglia modification: a randomized study. Heart Rhythm. 2011 May;8(5):672-8. doi: 10.1016/j.hrthm.2010.12.047. Epub 2010 Dec 31. PMID 21199686
- [Background] Edgerton JR, Brinkman WT, Weaver T, Prince SL, Culica D, Herbert MA, Mack MJ. Pulmonary vein isolation and autonomic denervation for the management of paroxysmal atrial fibrillation by a minimally invasive surgical approach. J Thorac Cardiovasc Surg. 2010 Oct;140(4):823-8. doi: 10.1016/j.jtcvs.2009.11.065. Epub 2010 Mar 17. PMID 20299028
- [Background] Yilmaz A, Geuzebroek GS, Van Putte BP, Boersma LV, Sonker U, De Bakker JM, Van Boven WJ. Completely thoracoscopic pulmonary vein isolation with ganglionic plexus ablation and left atrial appendage amputation for treatment of atrial fibrillation. Eur J Cardiothorac Surg. 2010 Sep;38(3):356-60. doi: 10.1016/j.ejcts.2010.01.058. Epub 2010 Mar 12. PMID 20227287
- [Background] Pokushalov E, Romanov A, Shugayev P, Artyomenko S, Shirokova N, Turov A, Katritsis DG. Selective ganglionated plexi ablation for paroxysmal atrial fibrillation. Heart Rhythm. 2009 Sep;6(9):1257-64. doi: 10.1016/j.hrthm.2009.05.018. Epub 2009 May 20. PMID 19656736
- [Background] Gelsomino S, Lozekoot P, La Meir M, Lorusso R, Luca F, Rostagno C, Renzulli A, Parise O, Matteucci F, Gensini GF, Crjins HJ, Maessen JG. Is ganglionated plexi ablation during Maze IV procedure beneficial for postoperative long-term stable sinus rhythm? Int J Cardiol. 2015 Aug 1;192:40-8. doi: 10.1016/j.ijcard.2015.04.259. Epub 2015 May 1. PMID 25985014